CLINICAL TRIAL: NCT06624787
Title: Development Of A Rapid Diagnostic Test To Identify Crimean-Congo Haemorrhagic Fever At The Point-Of-Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Medical Research Council (Other Government); MEDEX (Other); Mologic Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LSTM 24-044
Record Dates: First submitted 2024-08-14; First posted 2024-10-03 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-08

CONDITIONS: Crimean-Congo Haemorrhagic Fever
Keywords: CCHF; Medical Device; Lateral Flow; Rapid Diagnostic Test; LFT; RDT
MeSH Terms: conditions — Hemorrhagic Fever, Crimean | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Intervention Model Description: A diagnostic evaluation study where each participant undergoes both reference testing and the diagnostic testing
Masking Description: Operators performing the RT-PCR will be unaware to the RDT results. This removes bias of the RT-PCR and RDT results. The results of the RDTs will not be shared with the participants and the healthcare staff will be trained to not use the results, as the RDT is not an approved device for CCHF diagnosis. Participants will follow the local standard of care of CCHF diagnosis and management which dependent on the MoH RT-PCR result.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Rapid Diagnostic Test — The Liverpool School of Tropical Medicine (LSTM) in collaboration with Global Access Diagnostics (GADx) have achieved the development of the first RDT to detect CCHF viral antigens with a sensitivity and specificity that exceeds the minimum recommendation in the WHO target product profile (TPP)of >80% and >90% for sensitivity and specificity respectively for minimal performance in pre-clinical studies. The RDT is not only faster providing a test result within 20 minutes, but is also substantially cheaper than RT-PCR, and simpler to perform. A predicted price per test of around $5, whereas the current price of the RT-PCR test ranges from $1,000 to $1,200 for 96 reactions. The RDT does not require refrigeration or require specialist personnel to undertake, and the only additional apparatus needed is a stopwatch to monitor running time.

SUMMARY:
The goal of this medical device diagnostic evaluation study is to determine if this novel lateral flow device can detect Crimean-Congo Hemorrhagic Fever (CCHF) at the point of care in secondary health care clinics in Turkey. The main outcome is to determine the sensitivity and specificity of the tests for CCHF in samples of whole blood, serum and capillary blood compared to a gold-standard of PCR for participants that present at 4 endemic sites secondary health care clinics in Turkey in 492 adults who are suspected to have been infected with CCHF. The study aims to hopes to achieve at least the minimum required sensitivity of 90 % and specificity of 80 % as required by the WHO.

ELIGIBILITY:
Inclusion Criteria:

Participants aged 18 years or older Suspected CCHF infection that requires a RT-PCR diagnosis and venous blood draw Willingness to comply with study procedures and consent to the study Presents at 1 of 4 listed sites

Exclusion Criteria:

* In the investigators opinion should not be enrolled onto study (e.g., medical prudence or capacity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity | From the date/time of blood draw of the first participant until all diagnostic results have been received (up to two weeks from blood draw)
  To determine the sensitivity and specificity of RDT tests for CCHF in samples of whole blood, serum and capillary blood compared to a gold-standard of PCR for participants that present at 4 endemic sites secondary health care clinics in Turkey.

SECONDARY OUTCOMES:
Usability of RDT via questionnaires answered by end users. | Once all questionnaires have been completed, and quality checked - this should occur upto a month after the last recruit
  To determine the ease of use of the RDT at the point of care in CCHF-endemic settings by end users answering a questionnaire designed with a 5-point Likert scale
To determine the most suitable matrices that have the minimum TPP as required by the WHO for RDTs for CCHF detection. | From the date/time of blood draw of the first participant until all diagnostic results and questionnaires have been received - this should be completed upto a month after the last recruit
  Using the sensitivity, specificity, ease-of-use questionnaires, Positive predictive value, Negative predictive value and accuracy of RDT in all matrices to determine the most suitable matrix(ices) at the end-user setting.
Using the PPV, NPV and accuracy of the RDT in all matrices. | From the date/time of blood draw of the first participant until all diagnostic results have been received (up to two weeks from first blood draw of database lock)
  To determine the Positive predictive value (PPV), Negative predictive value (NPV) and Accuracy of the RDT in all matrices.
To determine the time taken for a CCHF result from blood draw. | From the date/time of blood draw of the first participant until all diagnostic results have been received (this should occur unto a month after the last recruit)
  Time from blood drawn to diagnostic result - (from upload to the MoH server, and from the site knowing the RT-PCR result)

OTHER OUTCOMES:
Exploratory Outcome 1 - To identify the types of clinical presentations in terms of SGS scores, symptomatic phases, and outcomes of CCHF in endemic areas of Turkey. | From the date/time of blood draw of the first participant until all diagnostic results and clinical information has been received - this should occur unto a month after the last recruit
  Sensitivity of the RDT among clinical, demographic, outcome subgroups of suspected CCHF-infected individuals in Turkey. Indirectly information of the clinical characteristics and demographics of the patients that require a CCHF diagnosis during 2025 CCHF in the selected clinics will be collected.
Exploratory Outcome 2 - Sensitivity of the RDT among local strains. Indirectly, information on the CCHFV strains circulating in Turkey during 2025 CCHF season will be collected. | From the date/time of blood draw of the first participant until all diagnostic results, clinical information and sequencing results have been received - this should occur upto 6 months after the last recruit
  Sequencing data on negative RDT results and PCR positive results to determine whether CCHFV strain has a negative impact on test sensitivity

IPD SHARING:
Plan to Share IPD: Undecided